CLINICAL TRIAL: NCT00065611
Title: Pulse Dexamethasone Over 48 Weeks for Podocyte Disease
Brief Title: Steroid Treatment for Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030226; 03-DK-0226
Record Dates: First submitted 2003-07-28; First posted 2003-07-29 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-09

CONDITIONS: Nephrosis; Focal Lipoid Glomerulosclerosis
Keywords: Steroids; Osteoporosis; Proteinuria; Minimal Change Disease; Focal Segmental Glomerulosclerosis; FSGS; MCD; Kidney Disease
MeSH Terms: conditions — Nephrosis; Osteoporosis; Proteinuria; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental; Macular dystrophy, corneal type 1; Kidney Diseases | interventions — Dexamethasone

INTERVENTIONS:
Drug: Oral dexamethasone — Stage I: Dexamethasone 25 mg/m2, 2 doses every 2 weeks over 48 weeks or dexamethasone 25 mg/m2, 4 doses every 4 weeks over 48 weeks.
  Stage II: 1.) Dexamethasone 50 mg/m2, 2 daily doses every 12 weeks, followed by 25 mg/m2, 2 daily doses every 2 weeks over 36 weeks, or 2.) Dexamethasone 50 mg/m2, 4 daily doses every 4 weeks over 12 weeks, followed by 25 mg/m2, 4 daily doses every 4 weeks over 36 weeks.
  over 36 weeks.

SUMMARY:
Focal segmental glomerulosclerosis (FSGS) and minimal change disease are kidney diseases that are associated with increased excretion of protein in the urine. Approximately half of FSGS patients will lose kidney function within 8 years of diagnosis and will require dialysis. The purpose of this study is to determine whether intermittent oral steroid therapy can cause sustained remission of FSGS and MCD.

Approximately 70 participants, including adults and children older than age 2, will be enrolled in this study. They will receive 48 doses of oral dexamethasone over a period of 48 weeks. One group will take two daily doses every 2 weeks; the other group will take four daily doses every 4 weeks. Doctors will monitor participants before, during, and after the steroid treatment with extensive exams and testing. At the completion of the study, researchers will evaluate the safety and efficacy of the drug treatment.

DETAILED DESCRIPTION:
The major causes of primary nephritic syndrome in adults and children are idiopathic podocyte diseases, minimal change (MCD) and focal segmental glomerulosclerosis (FSGS). Our objective is to determine whether intermittent oral dexamethasone administered over 48 weeks can induce complete remission in these patients. This is an open-label multi-center pilot study designed to obtain preliminary evidence of efficacy and to establish safety. This is part of a long-term effort to define the most effective mode of administering pulse dexamethasone and is expected to lead to a trial comparing daily prednisone to pulse dexamethasone.

We will enroll up to 70 patients with nephritic-level proteinuria due to biopsy-proven MCD (up to 30 patients) or FSGS (up to 40 patients). We will include adults and children greater than 2.0 years of age. Children with MCD must have received a minimum of 4 weeks and a maximum of 10 weeks of high-dose daily steroids, since many children are responsive to short courses of daily steroids; these requirements will define a steroid-resistant population. For children with FSGS and adults with MCD or FSGS, there is no minimum duration of prior steroids and there is a maximum of 8 weeks of prior high-dose daily steroids; these requirements will define a population that has received a short steroid course without response. If steroids have been used, inclusion criteria require persistent nephrotic syndrome (thus excluding steroid-sensitive nephrotic syndrome, whether steroid-dependent or frequently relapsing).

Patients may enroll at NIH or at collaborating centers. Those patients who enroll at NIH will visit the NIH Clinical Center at least 4 times. Patients enrolled at collaborating centers have the option to come to the NIH Clinical Center to complete research tests; under these circumstances they will be enrolled as NIH research subjects.

Patients will receive 48 doses of oral dexamethasone over a period of 48 weeks. Patients will be randomized to one of two arms: 2 daily doses every 2 weeks or 4 daily doses every 4 weeks. The rationale is to test whether increased frequency dosing has greater efficacy with acceptable safety. For adult patients, we have a record of safety with pulse dexamethasone from the FSGS Dexamethasone study as well as from published studies for other diseases. Therefore, for adults each pulse will be 50 mg/m(2) during the first 12 weeks and each pulse will be 25 mg/m(2) during the next 36 weeks. The trial for pediatric patients involves dose escalation, as there is little experience with pulse dexamethasone for podocyte diseases in this age group. In pediatric stage 1, each dexamethasone pulse will be 25 mg/m(2) over 48 weeks. When 4 patients in each arm have completed 48 weeks of therapy, safety and efficacy will be evaluated. If the evaluation is positive, we will embark on pediatric stage 2, in which dexamethasone pulses will be 50 mg/m(2) during the first 12 weeks and 25 mg/m(2) during the next 36 weeks (the same as the adult regimen).

The primary endpoint will be the presence of complete remission 48 weeks after beginning therapy. Secondary endpoints will include complete and partial remission at 48 weeks, and complete and partial remission at 104 weeks. Assessment of remission will be by 24 hour urine collection in adults and children greater than 13.0 years and first void urine samples in children less than 13.0 years. Patients will be evaluated for manifestations of steroid toxicity, including growth rate (children), ophthalmologic complications, adrenal suppression, osteoporosis, a vascular necrosis, and psychological disturbances.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults and children greater than 2.0 years of age are eligible. We will exclude children less than 2.0 years of age in light of the higher risk of steroid therapy in this age group and the higher likelihood genetic or syndromic FSGS, which is less likely to respond to steroids.
  2. Diagnosis:

     A) Biopsy-proven MCD and its variants, including IgM nephropathy and MCD with mesangial hypertrophy.

     B) Biopsy-proven FSGS, including idiopathic FSGS and collapsing FSGS. We will exclude patients with HIV-associated FSGS, as the risks of steroids are increased in these patients. We will exclude hyperfiltration FSGS associated with morbid obesity (BMI greater than 40 kg/m(2)), sickle cell anemia, reflux nephropathy, chronic tubular injury, congenital renal anomalies, and reduced nephron mass; the rationale is that these FSGS variants are considered refractory to steroids.
  3. Proteinuria: patients must have nephrotic range proteinuria. Baseline tests will be obtained when patients have been off all immunosuppressive therapy for greater than or equal to 1 month.
  4. Renal function: estimated GFR must be greater than or equal to 40 ml/min/1.73m(2) at the time of study entry; In children weighing less than 40kg, GFR will be estimated by the Schwartz formula and expressed as GFR/1.73m(2): GFR equal to [0.7 (males) or 0.57 (females) X height (cm)]/ serum creatinine.
  5. Angiotensin antagonists: Patients must be receiving angiotensin antagonist therapy, at any dose approved by the FDA. Nephrotic range proteinuria will be defined as urine protein greater than or equal to 3.5 g/1.73m(2)/d (adults) and greater than 50 mg/kg (children less than 40 kg) while receiving maximally tolerated dose of angiotensin antagonist therapy for at least 4 weeks prior to study entry.
  6. Prior immunosuppressive therapy:

     For children with MCD, we require a minimum of 4 weeks and a maximum of 10 weeks of daily steroid therapy at a dose of greater than or equal to 60 mg/m(2) with proteinuria persisting in the nephrotic range (excluding steroid-sensitive, steroid-dependent and frequently relapsing MDC).

     For children with FSGS and adults with MCD and FSGS, we require no minimum and a maximum of 8 weeks of daily or alternate day steroids at a dose of greater than 0.5 mg/kg with proteinuria persisting in the nephrotic range.

     Patients with prior immunosuppressive therapy other than steroids are eligible.
  7. If hypertensive, adequate blood pressure control (target BP less than 125/75 mm Hg at greater than 75% of measurements in adults).
  8. Women with reproductive potential who are sexually active must maintain an effective birth control regimen (oral contraceptive, intrauterine device, or barrier method plus spermicide) and must have a negative urine HCG test prior to beginning therapy.
  9. Patients must either have a negative PPD test within 3 months of study entry while off immunosuppressive therapy or, if they have a history of positive PPD, they must have appropriate evaluation to exclude untreated tuberculosis (with the advice of an Infectious Disease consultant).

EXCLUSION CRITERIA:

1. Patients with diabetes mellitus type 1 will be excluded, as these patients typically have brittle diabetic control that increases the risk of steroid treatment. Patients with diabetes mellitus type 2 will be included they manifest good glycemic control (glycosylated hemoglobin less than 7.5%), if they have lack proliferative retinopathy (the presence of proliferative retinopathy would place them at high risk for vision loss if steroids worsened glycemic control) and if they have had a renal biopsy within 6 months of study entry that shows no evidence for diabetic nephropathy.
2. Poorly controlled hypertension (greater than 25% of values greater than 125/75).
3. Evidence of significant chronic or occult infection. Specifically, subjects must not have evidence of active hepatitis B or hepatitis C infection, or HIV-1 infection, or untreated mycobacterial infection. Minor infections, such as skin or nail fungal infections or other infections with the advice of an Infectious Disease consultant, will not be the basis for exclusion.
4. Immunosuppressive medication other than glucocorticoids, whether for podocyte disease or another indication, must have been discontinued greater than 8 weeks prior to study entry. This does not apply to topical immunosuppressant medication.
5. Pregnancy.
6. Existence of any other condition that would complicate the implementation or interpretation of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adhikari M, Bhimma R, Coovadia HM. Intensive pulse therapies for focal glomerulosclerosis in South African children. Pediatr Nephrol. 1997 Aug;11(4):423-8. doi: 10.1007/s004670050309. PMID 9260238
- [Background] Yorgin PD, Krasher J, Al-Uzri AY. Pulse methylprednisolone treatment of idiopathic steroid-resistant nephrotic syndrome. Pediatr Nephrol. 2001 Mar;16(3):245-50. doi: 10.1007/s004670000494. PMID 11322372
- [Background] Houser MT, Jahn MF, Kobayashi A, Walburn J. Assessment of urinary protein excretion in the adolescent: effect of body position and exercise. J Pediatr. 1986 Sep;109(3):556-61. doi: 10.1016/s0022-3476(86)80143-3. PMID 3746552
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-DK-0226.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 patients were enrolled in the study, 4 of them are randomized to 2 dose every 2 week arm and 4 of them are randomized to 4 dose every 4 week arm.
Groups:
- 2 Doses Every 2 Weeks Arm: Patients in this arm receive 2 doses every 2 weeks
- 4 Doses Every 4 Weeks Arm: Patients in this arm receive 4 doses every 4 weeks
Period: Overall Study
Arm/Group | 2 Doses Every 2 Weeks Arm | 4 Doses Every 4 Weeks Arm
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Doses Every 2 Weeks Arm | 4 Doses Every 4 Weeks Arm | Total
Number analyzed (Participants) | 4 | 3 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (9) | 30 (5) | 35 (8) [31 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1 | 1 | 2
  African American | 2 | 2 | 4
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
Urine Protein [Mean (Standard Deviation); unit: g/d] | 11.2 (7.0) | 10.0 (1.9) | 10.8 (5.1)
CKD-EPI eGFR [Mean (Standard Deviation); unit: ml/min/1.73m^2] — estimate glomerular filtration rate (GFR) using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula
  ml/min/1.73m^2 | 59.2 (13.4) | 76.3 (21.4) | 66.6 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Remission Status of Patients After Intermittent Oral Dexamethasone Administered Over 48 Weeks
Description: Complete remission is defined as proteinuria <0.3 g/d. Partial remission is defined as a 50% fall in proteinuria compared to baseline, proteinuria <3.5 g/d, and a preserved estimated glomerular filtration rate (eGFR), specified as >60% of baseline. Limited response is defined as a 50% fall in proteinuria compared to baseline. All other outcomes are described as non-response.
Time Frame: 48 weeks from baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | 2 Doses Every 2 Weeks Arm | 4 Doses Every 4 Weeks Arm
Number analyzed (Participants) | 4 | 3
participants
  Limited response | 1 | 1
  Non-response | 2 | 1
  Partial remission | 1 | 1
  Complete remission | 0 | 0
Statistical Analysis 1: Comparison: 2 Doses Every 2 Weeks Arm vs 4 Doses Every 4 Weeks Arm; Test type: Superiority or Other; p = 0.9074, Chi-squared

2. Secondary Outcome: Urine Protein
Time Frame: 48 weeks from baseline
Measure: Mean (Standard Deviation); unit: g/d
Arm/Group | 2 Doses Every 2 Weeks Arm | 4 Doses Every 4 Weeks Arm
Number analyzed (Participants) | 4 | 3
g/d | 3.6 (0.7) | 6.2 (4.8)
Statistical Analysis 1: Comparison: 2 Doses Every 2 Weeks Arm vs 4 Doses Every 4 Weeks Arm; Test type: Superiority or Other; p = 0.4566, ANOVA

3. Secondary Outcome: CKD-EPI eGFR
Description: Estimate glomerular filtration rate (eGFR) using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula.
Time Frame: 48 weeks from baseline
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | 2 Doses Every 2 Weeks Arm | 4 Doses Every 4 Weeks Arm
Number analyzed (Participants) | 4 | 3
ml/min/1.73m^2 | 60 (16) | 73 (20)
Statistical Analysis 1: Comparison: 2 Doses Every 2 Weeks Arm vs 4 Doses Every 4 Weeks Arm; Test type: Superiority or Other; p = 0.3792, ANOVA

ADVERSE EVENTS:
Arm/Group | 2 Doses Every 2 Weeks Arm | 4 Doses Every 4 Weeks Arm
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/4
Other Adverse Events (participants affected / at risk) | 3/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Doses Every 2 Weeks Arm (N=4) | 4 Doses Every 4 Weeks Arm (N=4)
Tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute appendicitis, increased intraocular pressure (Gastrointestinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Doses Every 2 Weeks Arm (N=4) | 4 Doses Every 4 Weeks Arm (N=4)
Headache (General disorders) | 1 (1) | 0 (0)
sleep disturbance (General disorders) | 1 (1) | 1 (1)
Mood swings (General disorders) | 2 (2) | 1 (1)
Change in appetite (General disorders) | 0 (0) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
Impaired glucose tolerance (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cushingoid appearance (General disorders) | 0 (0) | 1 (1)
Muscle pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes